CLINICAL TRIAL: NCT03528811
Title: Evaluation of Microcirculation of Peripheral Vascular Disease in Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Maoquan Li, Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4250085-34
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Vascular Disease in Diabetes
Keywords: Diabetes; Peripheral Vascular Disease; Microcirculation
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Five points test of Tongji university (Other): We established the evaluatation and follow-up system of diabetes vascular disease based on the method called "Five points test of Tongji university" .
  Interventions: Diagnostic Test: Five points test of Tongji university

INTERVENTIONS:
Diagnostic Test: Five points test of Tongji university — In each group, we will evaluate the microcirculation of diabetic foot using the newly-established "Five points test of Tongji university" before or after the operation, and then compare the temperature of the five points with the other data.

SUMMARY:
The main aim of the present study was to evaluate the microcirculation of peripheral vascular disease in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with Peripheral vascular disease with or without diabetes. 2.Rutherford class 2-6. 3.Target lesions with a diameter reduction of at least 50% on angiography, and without past history of any intervention.

  4.Target vessel with 2.0--10.0mm in diameter and having a lesion of about 4cm-20cm in length.

  5.Written informed consent signed by the patients or representatives

Exclusion Criteria:

* 1.Previous bypass surgery or stent placement at the ipsilateral lower limb 2.History of intolerance to antiplatelet therapy, heparin, or contrast media. 3.Bleeding diathesis; 4.Active systemic bacterial infection; 5.Severely impaired renal function (serum creatinine level > 2.5 mg/dL. Expected survival time of less than 24 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Coincidence rate of "5 points test of Tongji university" | 12 months
  The primary study endpoint was that the coincidence rate of evaluating the microcirculation by the newly-established "5 points test of Tongji university" attains over 95% before and after operations as assessed by digital substraction angiography (DSA).

CONTACTS AND LOCATIONS:
Overall Officials: Xue Li, Ph.D, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tong ji University, Shanghai, China